CLINICAL TRIAL: NCT05864560
Title: Ankura™ AAA, Cuff and AUI Stent Graft System Post-Market Clinical Follow-Up: A Multi-center, Prospective, Single-arm, Open-label, Post-market Study
Brief Title: Ankura™ AAA, Cuff and AUI Stent Graft System Post-Market Clinical Follow-Up
Status: Active, not recruiting | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LT/TS/12C-2021-02
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Lifetech; Ankura; Endovascular Aneurysm Repair; Abdominal Aortic Aneurysm; Stent Graft System; EVAR; AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AAA Subjects: Patient diagnosed with Abdominal Aortic Aneurysm, who needs endovascular aortic repair.
  Interventions: Device: Ankura™ AAA Stent Graft System; Ankura™ Cuff Stent Graft System; Ankura™ AUI Stent Graft System

INTERVENTIONS:
Device: Ankura™ AAA Stent Graft System; Ankura™ Cuff Stent Graft System; Ankura™ AUI Stent Graft System — Patients will be implanted with Ankura™ AAA, Cuff or AUI Stent Graft System in accordance with the Instructions for Use (IFU).

SUMMARY:
The objective of the study is to collect real-world data on patient outcomes and evaluate the safety and performance of the Lifetech Ankura™ AAA Stent Graft System, Ankura™ Cuff Stent Graft System, Ankura™ AUI Stent Graft System and ZoeTrack™ Super Stiff Guidewire.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) is the most common true arterial aneurysm. Surgical management options for AAA include traditional Open Surgical Repair (OSR) and minimally invasive Endovascular Aneurysm Repair (EVAR). Multiple endovascular devices are commercially available for repair of AAA. Currently available endovascular grafts for infrarenal aortic repair share a bifurcated, modular design. Ankura™ Stent Graft Systems are minimally invasive endovascular devices that offer an alternative treatment for patients with AAA, which have been marketed worldwide for many years. In order to evaluate the long-term safety and performance of the investigational device from real world, this post-market clinical follow-up study is planned under the Regulation (EU) 2017/745. The study intends to enroll 162 subjects. The anticipated enrollment period is approximately 1.5 years and subjects will be followed for 3 years (36 months) post-implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with Abdominal Aortic Aneurysm (AAA), who needs endovascular aortic repair;
2. Patient's anatomy suits Ankura™ AAA and Cuff Stent Graft Systems, or AUI Stent Graft IFU requirements, which indicated by the following:

   1. Adequate iliac/femoral access vessel that is compatible with the required delivery system.
   2. Non-aneurysmal proximal aortic neck length ≥15mm.
   3. Non-aneurysmal proximal aortic neck diameter of 18-32mm.
   4. Proximal aortic neck angulation ≤ 60°.
   5. Distal iliac artery anchorage zone ≥15mm.
   6. Distal iliac artery diameter of i. 8-22 mm (for Ankura™ AAA and Cuff Stent Graft Systems), OR ii. 10-16 mm (for Ankura™ AUI Stent Graft System).
   7. Morphology suitable for endovascular repair.
3. Patient could understand the purpose of the clinical trial, agrees to comply with the requirements of the study including the 3-year follow-up, and signed the patient informed consent, will participate in the study.

Exclusion Criteria:

1. Age<18 years or Age>85 years;
2. Patients' life expectancy < 1 year;
3. Pregnant or plan to be pregnant or breast feeding;
4. Patient with any contraindications mentioned in the Ankura™ AAA and Cuff Stent Graft Systems, or in Ankura™ AUI Stent Graft system IFU:

   1. Patient with acute systemic infection;
   2. Patient with mesenteric blood flow mainly supplied by the inferior mesenteric artery;
   3. Patient with accessory renal artery original from abdominal artery;
   4. Patient who has allergic reaction to the device;
   5. Patient who is not suitable for endovascular repair in vascular morphology;
   6. Patient who cannot tolerate contrast agents due to renal insufficiency;
   7. Patient who is allergic to contrast agent;
   8. Patient's aneurysms neck has thrombus;
   9. Non-aneurysmal proximal aortic neck length <15mm;
   10. Non-aneurysmal proximal aortic neck diameter <18mm or >32mm;
   11. Proximal aortic neck angulation > 60°;
   12. Distal iliac artery anchorage zone <15mm;
   13. Distal iliac artery diameter: i. For Ankura™ AAA and Cuff Stent Graft Systems: <8mm or >22mm, OR ii. For Ankura™ AUI Stent Graft system: <10mm or >16mm.
5. Patient with traumatic aortic injury;
6. Patient with uncorrectable coagulopathy;
7. Patient with hereditary connective tissue disease, including but not limited to Marfan Syndrome or Ehlers-Danlos Syndrome;
8. Patient with concomitant thoracic aortic or thoraco-abdominal aneurysms；
9. Patient who weighs greater than 350 pounds (150kg) or cannot undergo accurate fluoroscopy examination due to obesity.
10. Acute myocardial infarction or heart failure (NYHA class III and IV), respiratory failure, malignant tumor and other serious systemic diseases.
11. Subject must not be participating in another study for an investigational drug and/or device that may clinically interfere with this study's endpoints.
12. Any condition (medical or anatomic) which makes the patient not suitable for endovascular repair according to the opinion of the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with Abdominal Aortic Aneurysm, who needs endovascular aortic repair.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Events (MAE) | within 30 days post-procedure
  MAEs are defined as all-cause death, myocardial infarction, renal failure, respiratory failure, paraplegia, stroke, and intestinal ischemia.
12-month Treatment Success Rate | 12 months post-procedure
  Rate of successful endovascular aneurysm repair with Ankura™ AAA and Cuff Stent Graft Systems or Ankura™ AUI Stent Graft system in 12 months. A successful repair should meet ALL the following requirements:
  1. Technical success, defined as delivery system delivered the stent graft at the desired position, stent graft deployed successfully.
  2. No aneurysm diameter dilation or aneurysm diameter dilation ≤ 5mm compared to baseline.
  3. No stent graft migration or stent graft migration ≤ 10mm.
  4. No re-intervention due to type I and III Endoleak.
  5. No aneurysm rupture.
  6. No conversion to Open Surgical Repair (OSR).
  7. No stent graft thrombosis.

SECONDARY OUTCOMES:
All-cause mortality | through 36 months post-procedure
Incidence of device-related or procedure-related SAE | through 36 months post-procedure
Incidence of abdominal aneurysm-related or stent graft-related secondary intervention, including Endovascular Aortic Repair (EVAR) and open surgery | through 36 months post-procedure
Incidence of stent migration (>10mm) | at 3-6 months, 12 months, and 24 months post-procedure
Incidence of stent fracture | at 3-6 months, 12 months, and 24 months post-procedure
Incidence of stent thrombosis | at 3-6 months, 12 months, and 24 months post-procedure
Incidence of stent embolization | through 36 months post-procedure
Immediate procedure success rate | immediately after the procedure
  Defined as Ankura™ stent graft is successfully implanted at the desirable place guided by Lifetech ZoeTrack™ Super Stiff Guidewire.
Incidence of Type I, III, IV Endoleak | at 3-6 months, 12 months, and 24 months post-procedure
Incidence of aneurysm enlargement (>5mm, compared to baseline) | at 3-6 months, 12 months and 24 months post-procedure
Incidence of aneurysm/vessel rupture | through 36 months post-procedure

CONTACTS AND LOCATIONS:
Locations (7):
- Bulgaria (2):
  - MBAL Heart and Brain EAD, Pleven
  - University Hospital for Active Treatment "Sofiamed", Sofia
- Greece (3):
  - Laiko - University Hospital of Athens, Athens
  - General University Hospital of Patras, Pátrai
  - Papageorgiou General Hospital, Thessaloniki
- Turkey (Türkiye) (2):
  - Ankara University Heart Center, Ankara
  - Ankara City Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No